CLINICAL TRIAL: NCT00633178
Title: Therapy for Prenatal Depression: Maternal & Fetal Effects
Brief Title: Effectiveness of Group Interpersonal Psychotherapy in Treating Women With Prenatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH072838, #4914; R34MH072838 (NIH)
Record Dates: First submitted 2008-03-07; First posted 2008-03-11 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2011-12

CONDITIONS: Depression
Keywords: Prenatal Depression; Postpartum Depression; Fetal Development; Interpersonal Therapy
MeSH Terms: conditions — Depression; Depression, Postpartum | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group Interpersonal Therapy (IPT) (Experimental): Participants will receive group interpersonal therapy.
  Interventions: Behavioral: Group interpersonal therapy (IPT)
- Treatment as Usual (ETAU) (Active Comparator): Participants will receive psychiatric treatment as usual.
  Interventions: Behavioral: Treatment as usual (TAU)
- No Treatment (No Intervention): Participants are healthy and will receive no treatment.

INTERVENTIONS:
Behavioral: Group interpersonal therapy (IPT) — Group IPT will include weekly treatment sessions with a psychiatrist for 12 weeks. The sessions will focus on overcoming relationship problems associated with depression. The first two and last sessions will be alone with the psychiatrist and the remaining sessions will be with a group of five to eight other pregnant women.
  Arms: Group Interpersonal Therapy (IPT)
Behavioral: Treatment as usual (TAU) — TAU will include referrals to outpatient treatment, which may include cognitive behavioral psychotherapy, insight-oriented psychotherapy, and/or antidepressant medication. TAU participants receiving psychotherapy will attend 12 weekly treatment sessions comparable to the IPT group sessions; treatment for TAU participants receiving medication for their depression may last longer than 12 weeks.
  Arms: Treatment as Usual (ETAU)

SUMMARY:
This study will evaluate the effectiveness of group interpersonal psychotherapy for preventing postpartum depression in pregnant women with depression and for improving healthy outcomes in their babies.

DETAILED DESCRIPTION:
The pregnancy and postpartum periods are times of remarkable emotional and physical change for a woman, making pregnant women more vulnerable to mood swings and depressive symptoms. It is estimated that approximately 10% to 15% of pregnant women experience depression, which can cause severe psychological distress for the woman as well as disturbances in infant development. Infants of depressed mothers are at a higher risk for developmental delays, behavioral problems, and difficulty eating and sleeping. Moreover, new data indicate that prenatal depression also may adversely affect brain development of the child even before birth. Despite the high prevalence rates of prenatal depression and its negative consequences, few studies have tested the effectiveness of interpersonal psychotherapy (IPT), a treatment for depression that focuses on interpersonal issues and relationships, during pregnancy. The administration of group prenatal IPT for depression may be effective in enhancing women's prenatal and postpartum moods and improving fetal and newborn functioning. This study will compare the effectiveness of group IPT with that of treatment as usual (TAU) for preventing postpartum depression in pregnant women with depression and for improving healthy outcomes in their babies. The study will also compare the fetal and newborn development of babies of healthy mothers with that of babies of depressed mothers.

This study will involve both healthy participants and participants with depression. All participants will start with an initial assessment visit between the 22nd and 23rd weeks of pregnancy. For participants who have shown signs of depression based on an initial phone interview, the initial visit will last about 2 hours and will include questions about medical and psychiatric history, depressive symptoms, and lifestyle habits and an examination of uterine blood flow using a Doppler ultrasound machine. Participants who do not show signs of depression will not undergo these assessments on the initial visit.

Participants found to be depressed on the first visit will then be assigned randomly to receive group IPT or TAU. Participants assigned to group IPT will attend 12 weekly psychiatrist-led sessions that will focus on overcoming relationship problems associated with depression. The first two and last sessions will be alone with the psychiatrist and the remaining sessions will be with a group of five to eight other pregnant women. Participants assigned to TAU will be referred to outpatient treatment, which may include cognitive behavioral psychotherapy, insight-oriented psychotherapy, and/or antidepressant medication. TAU participants receiving psychotherapy will attend 12 weekly treatment sessions comparable to the IPT group sessions; treatment for TAU participants receiving antidepressant medication may last longer than 12 weeks. During the treatment period, all participants will fill out weekly forms about their moods and will have monthly interviews with a psychiatrist. Upon completion of treatment, participants will have a 30-minute final evaluation meeting.

All participants, including healthy participants, will be asked to attend two sessions focused on their babies' development, one occurring between the 36th and 38th weeks of pregnancy and one shortly after giving birth. During the first developmental session, participants will complete a questionnaire about mood; undergo heart rate, breathing, and blood pressure monitoring; undergo an ultrasound; and perform a word matching task. The second developmental session will occur between 20 and 30 hours after birth of the baby and will include a newborn testing session that will consist of physiological and neurobehavioral assessments. Healthy participants' study participation will be over upon completion of the second developmental session. Depressed participants will be contacted by phone once every 2 weeks for 6 months after giving birth.

ELIGIBILITY:
Inclusion Criteria:

* Score of at least 10 on the Edinburgh Postnatal Depression Scale (EPDS)

Exclusion Criteria:

* Multi-fetal pregnancy
* Taking medications that affect the cardiovascular system (e.g., doxazosin)
* History of suicide attempt or current suicidal ideation
* Psychotic features
* Life-time history of bipolar disorder
* Current eating disorder
* Currently diagnosed with any of the following: obsessive compulsive disorder, major depression with melancholic features, severe major depression, panic disorder, organic brain syndrome, mental retardation, antisocial personality disorder, borderline personality disorder, or presence of three or more schizotypal features
* Smokes cigarettes
* Substance dependence or abuse
* Complicated pregnancy or delivery
* Premature delivery
* Neonate medical/developmental problems
* Taking a psychotropic medication at the time of the initial phone contact with study investigators

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2005-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Improved prenatal mood | Measured during the prenatal period (pregnant participants enroll at 23/24 weeks gestation and are assessed through 40 weeks of gestations)
  Hamilton Scales for Depression Score
Postpartum depression | Measured during the postpartum period (pregnant participants enroll at 23/24 weeks gestation and are assessed through 40 weeks of gestations)
  Hamilton Scales for Depression Score

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Monk, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States